CLINICAL TRIAL: NCT03346590
Title: Evolution of Total Energy Expenditure and Its Various Components in Active Rheumatoid Arthritis (RA)Treated With Anti-TNF Agents and Comparison With Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-365; 2017-A01654-49 (Other: 2017-A01654-49)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Active Rheumatoid Arthritis

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16 patients with active RA (Active Comparator): Women over 18 years old with proven active (DAS28 >3.2) RA, diagnosed based on ACR/EULAR 2010 criteria, receiving biological anti-TNF treatment for the first time.
  Covered by social security. Capable of giving informed consent and acceding to the requirements of the study. For high-resolution echocardiography: no hypertension, diabetes or history of cardiovascular disorders.
  Interventions: Behavioral: Energy metabolism of patients suffering from RA
- 8 Healthy volunteers (control group) (Sham Comparator): Healthy volunteers (control group) The healthy female controls will be enrolled from the Centre de Recherche en Nutrition Humaine (CRNH) list of volunteers and matched to the RA patients according to age ±5 years and BMI class (<25; 25-30; >30).
  Interventions: Behavioral: Energy metabolism of patients suffering from RA

INTERVENTIONS:
Behavioral: Energy metabolism of patients suffering from RA — Energy metabolism of patients suffering from RA

SUMMARY:
Chronic inflammation in rheumatoid arthritis is associated with adiposity, sarcopenia, cachexia, reduced activity due to functional impairment, and anti-inflammatory drugs. Patients frequently gain weight when taking anti-tumor necrosis factor (TNF) medication, prompting questions about the underlying mechanism and long-term cardiovascular and metabolic tolerance associated with these drugs The primary objective of this study is to analyze the impact of anti-TNF treatment during the first year of administration on the energy metabolism of patients suffering from RA, assessed as an absolute value (before-after) and in comparison with a standard measured in healthy matched subjects.

DETAILED DESCRIPTION:
Few studies have been focused on the combined evolution of body composition, energy expenditure, physical activity, muscle performance, and nutritional intake in patients taking anti-TNFs.

This study's objective is to assess the impact of anti-TNF treatment during the first year of administration on the energy metabolism of RA patients, measuring variations in basal daily energy expenditure and per type of expenditure using indirect calorimetry with calorimetric chambers. Investigator also aim to define standardized values for RA patients compared to healthy matched controls and to be able to monitor the evolution of these different values during treatment compared to this standard.

This will be an exploratory study with a longitudinal follow-up of the cohort in patients treated in a market authorization context and involving a case/control study. Investigator judged the inclusion of healthy controls justified by the current lack of data comparing the different components of energy metabolism in active RA patients versus healthy subjects using calorimetric chamber measurement. The aim is to obtain reference values to situate RA-specific values in comparison before and after treatment. Investigator considered selecting controls from the RA patients unjustified given how essential it is to commence treatment in active RA cases (1 year with placebo not justifiable). A previously-treated inactive RA population with no inflammation would not be comparable to patients with active RA, and neither would a population with active RA treated with conventional treatment or a different biotherapy to anti-TNFs. Investigator also chose to perform a second assessment at 6 months without calorimetric chamber measurement but rather an indirect measurement using actimetry in order to limit costs and patients lost-to-follow-up due to treatment modification (failure or intolerance), all the while maintaining full assessment at 12 months. Scheduling the assessment at 12 months is justified by published studies' reports of delay before significant weight gain manifests, and enables us to maintain homogeneity as regards variations in physical activity and nutritional intake linked to seasonal changes.

ELIGIBILITY:
Inclusion Criteria:

* RA patients Women over 18 years old with proven active (DAS28 >3.2) RA, diagnosed based on ACR/EULAR 2010 criteria, receiving biological anti-TNF treatment for the first time.

Covered by social security. Capable of giving informed consent and acceding to the requirements of the study.

For high-resolution echocardiography: no hypertension, diabetes or history of cardiovascular disorders.

- Healthy volunteers (control group) The healthy female controls will be enrolled from the Centre de Recherche en Nutrition Humaine (CRNH) list of volunteers and matched to the RA patients according to age ±5 years and BMI class (<25; 25-30; >30).

Exclusion Criteria:

* Refusal to sign consent form.

  * Patients under guardianship or curatorship.
  * Previous exposure to biological treatment in the course of their disease.
  * Suffering from a condition potentially influencing energy metabolism: infection, cancer, diabetes, thyroid dysfunction, psychiatric disorder, current smoker, pregnancy.
  * High physical activity level, based on short-form IPAQ questionnaire.
  * Variations in weight exceeding 5% of body weight in the previous 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Continuous measurement of energy expenditure and cardiac rhythm in calorimetric chamber | for 36 hours
  Continuous measurement of energy expenditure and cardiac rhythm in calorimetric chamber for 36 hours: at rest, waking, during two physical activity sessions (treadmill walking at 4km/h for 30min), sleeping.
Indirect assessment of energy expenditure | for 4 days
  Indirect assessment of energy expenditure by measuring physical activity using home actimetry(Armband) under normal living conditions for 4 days and in the calorimetric chamber for calibration.
Nutritionist assessment of nutritional intake | during the 2 days preceding energy expenditure measurement.
  Nutritionist assessment of nutritional intake during the 2 days preceding energy expenditure measurement.
Previously-scheduled tests for the RCVRIC protocol | at day 1

SECONDARY OUTCOMES:
Indirect assessment of energy expenditure via measurement of physical activity using calibrated actimetry (Armband) | at 6 months
  Indirect assessment of energy expenditure via measurement of physical activity using calibrated actimetry (Armband) at home in normal living conditions over 4 days.
Nutritionist evaluation of nutritional intake over 2 days | at 6 months
Previously-scheduled tests for the RCVRIC study protocol (M6): | at 6 months
  DXA, pQCT, physical strength and performance, physical activity and nutrition questionnaires, cardiovascular risk, serum and urine bank research.

CONTACTS AND LOCATIONS:
Overall Officials: Anne TOURNADRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France